CLINICAL TRIAL: NCT05457465
Title: Assessing the Impact of Cannabidiol for Anxiety and Depression in Bipolar Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Staci Gruber, Ph.D., Director, Marijuana Investigations for Neuroscientific Discovery; Director, Cognitive and Clinical Neuroimaging Core, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000825
Record Dates: First submitted 2022-06-21; First posted 2022-07-14 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Disorder
Keywords: Cannabidiol
MeSH Terms: conditions — Bipolar Disorder | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hemp-Derived Cannabidiol Solution (Experimental): Patients will administer a custom-formulated, hemp-derived, high-CBD solution twice daily for 4 weeks
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Custom formulation of a hemp-derived, high-CBD product that contains no THC.

SUMMARY:
Preliminary data have suggested that cannabidiol (CBD) may have a number of clinical benefits, including anti-anxiety and antidepressant properties. This study is a pilot open-label clinical trial assessing a custom-formulated high-CBD product over the course of 4 weeks in patients with bipolar disorder who experience anxiety.

DETAILED DESCRIPTION:
This investigation will be the first of its kind to conduct a clinical trial of an industrial hemp-derived high-CBD product in individuals with bipolar disorder who experience anxiety. Despite the recent interest in medical cannabis and cannabinoid-based products, the availability of hemp-derived products in all 50 states, and preliminary and anecdotal evidence suggesting that hemp-derived products may have a profound anxiolytic effect, along with potential antidepressant effects, no studies have conducted a clinical trial of a hemp-derived product in individuals with bipolar disorder who suffer from anxiety.

This investigation consists of a four-week open-label clinical trial of the custom formulated hemp-derived high-CBD solution. Participants will be pre-screened by phone in order to evaluate their eligibility for the study. If approved, potentially eligible participants will come to the hospital for a screening visit, and will complete a structured clinical interview, clinical and quality of life questionnaires, a urine screen, and a blood draw. Eligible participants will return for a baseline visit consisting of additional clinical and quality of life questionnaires, a brief cognitive assessment, and a buccal swab for genetic analysis. Participants will be given study product to use for the duration of the study, and will be instructed to self-administer the solution under the tongue twice daily for four weeks. Throughout the treatment period, participants will complete short in-person or remote visits on a weekly basis, where they will complete questionnaires about their mood and quality of life. Participants will also return to the hospital for a final visit after four weeks of treatment to complete additional questionnaires and cognitive assessments.

ELIGIBILITY:
Inclusion Criteria:

* Provides informed consent
* Between the ages of 18-65
* Fluent in English
* Meets DSM-5 criteria for bipolar disorder (type I or II)
* Experiences at least moderate levels of anxiety (as evidenced by self-reported rating scales)
* On a stable pharmacotherapeutic regimen

Exclusion Criteria:

* Not fluent in English
* Estimated IQ <75
* Current substance use disorder, current eating disorder, current or past psychotic disorder (e.g. schizophrenia, schizoaffective disorder)
* Endorsement of suicidality
* Experiencing acute manic episode
* Experiencing acute depressive episode
* History of head injury/loss of consciousness >5 minutes
* Current regular use of cannabinoid products
* Pregnant or breastfeeding
* Presence of serious medical illness or neurological disorder
* Allergy to palm oil
* Current use of valproate or divalproex; other concomitant medications may result in exclusion on a case-by-case basis
* Currently enrolled in another clinical trial that involves a treatment
* Elevated LFTs at screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported ratings of anxiety on the Beck Anxiety Inventory (BAI) | 4 weeks
  Anxiety will be assessed using a number of self-report and administered clinical ratings scales: the primary outcome measure will be the Beck Anxiety Inventory (BAI), which is a 21-item self-report measure used to rate subjective, somatic, and panic-related symptoms of anxiety on a scale of 0 (not at all) to 3 (severely). The total score ranges from 0 (no anxiety) to 63 (severe anxiety).

SECONDARY OUTCOMES:
Change in self-reported ratings of depression on the Beck Depression Inventory (BDI) | 4 weeks
  Depressive symptoms will be assessed using the Beck Depression Inventory (BDI), which is a 21-item self-report measure used to rate symptoms of depression on a scale of 0 (none) to 3 (very much). The total score ranges from 0 (no depressive symptoms) to 63 (severe depressive symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided